TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

### STATISTICAL ANALYSIS PLAN

### **Protocol TT-018**

A Phase 1/2a Study to Determine the Dose Response Pharmacokinetics of TSX-011 (Testosterone Undecanoate) in Hypogonadal Males

**PAREXEL Study Number 235004** 

Version: Final 1.0 Date: 13 June 2018

TesoRx Pharma, LLC Protocol Number TT-018 Final 1.0 13 June 2018

### SIGNATURE PAGE - TESORX PHARMA

### **Declaration**

The undersigned agree to the statistical analyses and methods described in this SAP.

Karl Begin / Date (dd mmm yyyy)
TesoRx Pharma, LLC

Michael Oefelein, MD, FACS TesoRx Pharma, LLC

Date (dd mmm yyyy)

21 June 2018

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

June 2018

Date (dd mmm yyyy)

### SIGNATURE PAGE - PAREXEL

### **Declaration**

The undersigned agree to the statistical analyses and procedures of this clinical study.

Prepared by: Walter Heber, MSc Associate Manager, EP Biostatistics

PAREXEL International Corporation

Page 3 of 84

TesoRx Pharma, LLC Protocol Number TT-018 Final 1.0 13 June 2018

### **TABLE OF CONTENTS**

| SIGNA | TURE PAGE – TESORX PHARMA | 2 |
|---------|--------------------------------------------------|----|
| SIGNA | TURE PAGE - PAREXEL | 3 |
| TABLE | E OF CONTENTS | 4 |
| 1. | STATISTICAL ANALYSIS PLAN | 9 |
| 2. | STUDY OBJECTIVES AND HYPOTHESES PER PROTOCOL | 9 |
| 2.1 | PRIMARY OBJECTIVES | 9 |
| 2.2 | SECONDARY OBJECTIVES | 9 |
| 2.3 | EXPLORATORY OBJECTIVES | 9 |
| 3. | STUDY DESIGN PER PROTOCOL | 10 |
| 3.1 | STUDY ENDPOINTS PER PROTOCOL | 12 |
| 3.2 | STUDY POPULATION | 13 |
| 3.3 | SAMPLE SIZE | 13 |
| 3.4 | RANDOMIZATION AND BLINDING | 13 |
| 3.5 | DOSE ADMINISTRATION | 13 |
| 3.5.1 | ADAPTIVE DESIGN CRITERIA | 15 |
| 3.5.1.1 | DOSE ADJUSTMENT PERIOD 3 DAY 16 | 15 |
| 3.5.1.2 | DOSE ADJUSTMENT PERIOD 3 DAY 26 | 16 |
| 3.6 | MEAL ADMINISTRATION | 18 |
| 3.7 | INTERIM ANALYSIS | 19 |
| 4. | PAREXEL STUDY ANALYSIS VARIABLES | 19 |
| 4.1 | DEMOGRAPHIC AND BACKGROUND VARIABLES | 19 |
| 4.2 | SAFETY VARIABLES | 19 |
| 4.2.1 | ADVERSE EVENTS | 19 |
| 4.2.2 | CLINICAL LABORATORY TESTS | 19 |
| 4.2.2.1 | OTHER LAB ASSESSMENTS - TESTOSTERONE LEVELS, PSA | 21 |
| 4.2.3 | VITAL SIGNS | 21 |
| 4.2.4 | ELECTROCARDIOGRAMS | 22 |
| 4.2.5 | PHYSICAL EXAMINATION | 22 |
| 4.2.6 | CONCOMITANT MEDICATIONS | 22 |
| 4.3 | QUALITY OF LIFE ASSESSMENTS | 23 |
| 4.4 | PHARMACOKINETIC VARIABLES | 23 |
| 4.4.1 | PHARMACOKINETIC PARAMETER CALCULATION METHODS | 25 |

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

| 4.5 | PHARMACODYNAMIC VARIABLES | 25 |
|---|---|---|
| 4.6 | EFFICACY VARIABLES | 25 |
| 4.7 | ANALYSIS POPULATIONS | 25 |
| 4.7.1 | SAFETY POPULATION | 25 |
| 4.7.2 | PHARMACOKINETIC POPULATION (PK) | 25 |
| 5. | STATISTICAL REPORTING | 26 |
| 5.1 | GENERAL CONSIDERATIONS FOR DATA PRESENTATIONS | 26 |
| 5.2 | TREATMENT IDENTIFICATION | 27 |
| 6. | SUBJECT AND TREATMENT INFORMATION | 27 |
| 6.1 | SUBJECT DISPOSITION | 27 |
| 6.2 | ELIGIBILITY CRITERIA AND PROTOCOL DEVIATIONS | 28 |
| 6.3 | EXCLUSION TESTS | 28 |
| 6.4 | DEMOGRAPHIC DATA | 28 |
| 6.5 | MEDICAL HISTORY | 28 |
| 6.6 | CONCOMITANT MEDICATION | 28 |
| 6.7 | DOSE ADMINISTRATION | 28 |
| 7. | PHARMACOKINETIC CONCENTRATIONS AND PARAMETERS | 29 |
| 7.1 | PLASMA CONCENTRATIONS | 29 |
| 8. | SAFETY ANALYSIS | 29 |
| 8.1 | ADVERSE EVENTS | 29 |
| 8.2 | CLINICAL SAFETY LABORATORY TESTS (HEMATOLOGY, CHEMISTRY, URINALYSIS) | 31 |
| 8.2.1 | HEMATOLOGY AND CHEMISTRY | 31 |
| 8.2.2 | URINALYSIS | 31 |
| 8.2.3 | LABORATORY COMMENTS | 32 |
| 8.2.4 | OTHER LABORATORY ASSESSMENTS | 32 |
| 8.3 | VITAL SIGNS | 32 |
| 8.4 | 12-LEAD SAFETY ECG | 32 |
| 8.5 | PHYSICAL EXAMINATION | 33 |
| 8.6 | IPSS QUESTIONNAIRE | 33 |
| 8.7 | QOL QUESTIONNAIRE | 33 |
| 9. | REPORTING OUTPUT | 34 |
| 10. | REFERENCES | 34 |
| 11. | SUMMARY TABLES | 35 |
| 12 | LISTINGS | 36 |

TesoRx Pharma, LLC

| Protocol Number TT-018 | | 13 June 2018 |
|------------------------|----------------|--------------|
| 13. | TABLE SHELLS | |
| 14 | LISTING SHELLS | 56 |

Final 1.0

TesoRx Pharma, LLC Final 1.0
Protocol Number TT-018 13 June 2018

#### **Abbreviations and Definitions**

AE Adverse event

ALT L-alanine aminotransferase AST L-aspartate aminotransferase

AUC Area under the curve

AUClast Area under the concentration versus time curve from time 0 to the last

measurable concentration

AUCt Area under the concentration versus time curve, from time 0 to the last

measurable concentration on or before time t

AUCinf Area under the concentration versus time curve from time 0 to infinity

BLQ Below the lower limit of quantification

BMI Body Mass Index BUN Blood urea nitrogen

Cavg,ss Steady-state average drug concentration

CI Confidence interval

CL/F Apparent total body clearance after oral dosing

CS Clinically significant

Cmax Maximum plasma TSX-011 concentration determined directly from the

concentration-time profile

Cmin Minimum drug concentration

CV Coefficient of variation CYP Cytochrome P450 DHT Dihydrotestosterone

DHTU Dihydrotestosterone undecanoate

ECG Electrocardiogram

HBsAg Hepatitis B surface antigen
HIV Human immunodeficiency virus
IMP Investigational Medicinal Product
Lambda z Apparent elimination rate constant

MedDRA Medical Dictionary for Regulatory Activities

NCS Not clinically significant

PDQ Psychosexual Daily Questionnaire

PK Pharmacokinetic
SAE Serious adverse event
SAP Statistical Analysis Plan
SD Standard deviation
SOC System Organ Class

t<sub>1/2</sub> Apparent elimination half-life
TEAE Treatment-emergent adverse event

Tmax Time of the maximum measured concentration over the specified

interval. If the maximum value occurs at more than one time point, Tmax

is defined as the first time point with this value.

Tmin Time of the minimum measured concentration over the specified interval

TesoRx Pharma, LLC Final 1.0
Protocol Number TT-018 13 June 2018

TU Testosterone undecanoate

Vss/F Volume of distribution at steady state after oral dosing

WHO World Health Organization

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

#### 1. Statistical Analysis Plan

This Statistical Analysis Plan (SAP) is based on the final protocol TT-018 dated 31 July 2017 and incorporates protocol Version 2.0 dated 26 October 2017 and Version 3.0. dated 05 March 2018. The SAP provides details on the planned statistical methodology for analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures. It describes the safety, pharmacokinetic (PK) variables, the anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP covers the planned analysis of all data collected electronically in Clinbase and provided by external vendors.

### 2. Study Objectives and Hypotheses per Protocol

### 2.1 Primary Objectives

To assess the pharmacokinetics (PK) of total testosterone after oral dosing of TSX-011 in hypogonadal adult male subjects following: 1) single ascending doses, and 2) single or multiple daily doses administered over a 30-day period in a fixed-dose and dose-adjustment adaptive design.

### 2.2 Secondary Objectives

- To assess the safety and tolerability of TSX-011 in hypogonadal adult male subjects by evaluating treatment-emergent adverse events (TEAEs).
- To assess the PK of free testosterone, testosterone undecanoate (TU), dihydrotestosterone (DHT), and dihydrotestosterone undecanoate (DHTU) after oral dosing of TSX-011 in hypogonadal adult male subjects following: 1) single ascending doses, and 2) single or multiple daily doses administered over a 30-day period in a fixed-dose and dose-adjustment adaptive design.

### 2.3 Exploratory Objectives

• To assess the effect of TSX-011 on hypogonadal symptoms as measured by hypogonadal quality of life (QOL) questionnaires: Aging Male Symptom (AMS) scale, Multinational Survey of the Aging Male-7 (MSAM-7; libido questions only), and Psychosexual Daily Questionnaire (PDQ).

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

• To determine the preferred method of PK specimen collection - Serum or enzyme inhibited plasma.

### 3. Study Design per Protocol

The study will be conducted as an open-label 3-period investigation as follows:

- Period 1. Ascending single-dose period: 190 mg TSX-011 (fed and fasted), 380 mg TSX-011 (fed), and 570 mg TSX-011 (fed).
- Period 2. 380 mg TSX-011 twice daily dosing period of 15 days in fed conditions.
- Period 3. Dose-adjusted adaptive design period: TSX-011 dose adjustment permitted on Day 16 and Day 26 based on 6 hours postdose (± 15 minutes) testosterone level on Day 8 and Day 19, respectively; dosing period of 15 days.

Dosing amounts of TSX-011 in this protocol refer to TU amounts.

Up to 24 subjects will be enrolled in this study to yield 16 evaluable subjects, and it is desired that the same 24 subjects participate in all 3 study periods.

The three initial cohorts of 3 subjects each will complete Periods 1, 2, and 3 prior to enrolment of remaining subjects. Interim review of safety and efficacy of TSX-011 will occur prior to enrolment of remaining subjects in the study. Dose response and optimum dosing conditions and PK specimen collection methods (serum vs. enzyme inhibited plasma) will be confirmed prior to remaining subject enrolment.

Enrolment will be managed to result in at least 10 evaluable native Japanese subjects. Subjects may be replaced at the discretion of the Sponsor in consultation with the Principal Investigator (PI).

A schematic of the study design is given in the below figure:

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

### **Study Design for Study TT-018**



TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

### 3.1 Study Endpoints per Protocol

The primary endpoints of the study are PK parameters for testosterone after TSX-011 administration under fed (or fasted [Period 1, 190 mg dose only]) conditions as described below:

- 1. Period 1 (ascending single doses):
  - a. Total (actual measured) testosterone, AUCt, Cmax, Tmax, Cmin, Tmin, and Cmax to Cmin ratio.
  - b. Baseline-corrected (BC) testosterone:  $\lambda z$ ,  $t^1/_2$ , CL/F,  $V_{ss}/F$ ,  $C_{max}$ , AUClast, and AUC $_{\infty}$ .
- 2. Period 2 (twice-daily dosing) Days 1 and 15 and Period 3 (dose-adjustment adaptive design) Day 30:
  - a. Total testosterone: AUCt, Css,avg, Cmax, Tmax, Cmin, Tmin, and Cmax to Cmin ratio.

The secondary endpoints of the study are as follows:

- 1. Number and severity of TEAEs and results of physical examinations, electrocardiograms (ECGs), vital sign measurements, and clinical laboratory tests (serum chemistry, hematology, and urinalysis) following a single dose of TSX-011 and following a single- or multiple-daily dose regimen of TSX-011 using a fixed-dose or a dose-adjustment adaptive design.
- 2. PK parameters (AUCt, Cmax, Tmax, Cmin, and Cavg) for free testosterone, TU, DHT, and DHTU under fed (or fasted [Period 1, 190 mg dose only]) conditions following: 1) ascending single doses of TSX-011, and 2) single- or multiple-daily dose regimen of TSX-011 using a fixed-dose and dose-adjustment adaptive design.

The exploratory endpoints of the study are as follows:

- 1. Hypogonadal symptoms as measured by the hypogonadal QOL questionnaires: AMS scale, MSAM-7 (libido questions only), and PDQ.
- 2. Duplicate PK analysis (serum and enzyme inhibited plasma) in the first 9 subjects enrolled.

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

### 3.2 Study Population

The study population will consist of hypogonadal adult male subjects 18 to 75 years of age at time of study enrolment. Subjects must be able to provide written informed consent and meet all the inclusion criteria and none of the exclusion criteria as stated in the protocol.

Hypogonadal males are those with at least 1 serum testosterone level <350 ng/dL, 10 am [ $\pm$  2 hour] sample taken during the screening period.

### 3.3 Sample Size

The study is a proof-of-concept study with adaptive dosing. The sample size chosen for this study was selected without statistical considerations but has been determined adequate to meet the study objectives.

### 3.4 Randomization and Blinding

This is a non-randomized study. All subjects will be exposed to the same set of treatment administrations and will be dosed in all periods using non-random assignment to treatment.

If Period 2 Day 8 (6 hours postdose  $\pm$  15 minutes) total testosterone is >800 ng/dL, subjects will be assigned by non-random assignment in a 1:1 ratio to receive:

- Schedule A: 317 mg (TU) TSX-011 twice daily OR
- Schedule B: 507 mg (TU) TSX-011 once daily

Period 2 subjects will be stratified during treatment assignment per their Japanese/non-Japanese classification.

Overall enrolment will be managed to result in at least 10 evaluable Japanese subjects.

All treatment assignments for all periods of dosing will be managed within the electronic data capture system. The study is an open-label study, and as such, no blinding will be performed.

#### 3.5 Dose Administration

The investigational product is TSX-011.

TSX-011 capsule(s) will be administered orally with at least 240 mL of water.

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

Dosing (swallowing capsules) should be completed within 5 minutes of starting. All drug administration procedures will be performed at the clinical study unit during confinement. The actual time of each dose administration will be recorded to the nearest minute, and this will be used in conjunction with the actual sample times to determine PK parameters as appropriate.

### Period 1

This is conducted as an ascending single-dose study of TSX-011 at 3 doses, with the lowest dose administered under fed and fasted conditions: 190 mg TSX-011 in the fed state, 190 mg TSX-011 in the fasted state, 380 mg TSX-011 in the fed state, and 570 mg TSX-011in the fed state. Before exposure to TSX-011, a 24-hour baseline measurement of testosterone and DHT will be performed for each subject. Samples for analysis of testosterone will be obtained at the following time points on Day -1: hour 0 (8 am  $\pm$  60 minutes) and 1.5, 3, 4.5, 6, 8, 12, 16, and 24 hours ( $\pm$  15 minutes for each time point). Day -1 is during screening (prior to initial dose). Day -1 endogenous blood samples are taken to establish pre-dosing T levels.

The day following the sampling for endogenous testosterone (Day 1) in Period 1, each subject will receive the first single dose of TSX-011 (190 mg) under fed conditions. Following administration of TSX-011, blood samples will be obtained over a 24-hour period for PK analysis. Subjects will undergo a minimum 3-day and up to 7-day washout period between each of the doses of TSX-011 in Period 1. After the 570 mg TSX-011 dose in Period 1, a minimum 3-day and up to 7-day (14 day for three initial 3 subject cohorts) washout period will occur before the start of Period 2.

### Period 2

Subjects in a fed state will receive 380 mg TSX-011 twice daily (8 am  $\pm$  60 minutes and 6 pm  $\pm$  60 minutes) for 15 days (Days 1 through 15). Pharmacokinetic assessments over 24 hours will occur on Days 1 and 15. On Day 8 in Period 2, before the morning dose, a trough PK blood sample will be drawn. In addition, on Day 8, 6 hours ( $\pm$  15 minutes) after the morning dose, testosterone levels will be obtained and used to dose adjust according to the adaptive dosing design described below. The TSX-011 dose will be adjusted up or down beginning with the Day 16 (Period 3) morning dose, based on established dosing rules described below.

### Period 3

Period 3 is a dose-adjusted adaptive design period that begins on Day 16, with the first adjusted TSX-011 dose administered in the fed state on a once-daily or twice-daily schedule. The 6-hour postdose (± 15 minutes) testosterone level on Day 19 will

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

be used to perform the second and final TSX-011 dose adjustment, based on established criteria.

As specified by the dose adjustment rules below, Day 26 begins with either a oncedaily, twice-daily, or thrice-daily fed dose schedule. The thrice-daily dose schedule will be administered only to non-responders (C<sub>avg</sub> testosterone <350 ng/dL despite 1 dose adjustment). On Day 30, a 24-hour PK assessment will be performed, and the subject's participation in the study is completed the morning of Day 31.

### 3.5.1 Adaptive Design Criteria

### 3.5.1.1 Dose Adjustment Period 3 Day 16

- If Period 2 Day 8 (6 hours postdose ± 15 minutes) total testosterone is <350 ng/dL, adjust the first dose of Period 3 (Day 16 dose) to 570 mg (TU) TSX-011 twice daily.
- If Period 2 Day 8 (6 hours postdose ± 15 minutes) total testosterone is ≥350 ng/dL and <500 ng/dL, adjust the first dose of Period 3 (Day 16 dose) to 443 mg (TU) TSX-011 twice daily.
- If Period 2 Day 8 (6 hours postdose ± 15 minutes) total testosterone is 500 to 800 ng/dL, inclusive, maintain first dose of Period 3 (Day 16 dose) at 380 mg (TU) TSX-011 twice daily.
- If Period 2 Day 8 (6 hours postdose ± 15 minutes) total testosterone is >800 ng/dL, the first dose in Period 3 (Day 16 dose) will be by manual assignment in a 1:1 ratio to receive either:
  - o Schedule A: 317 mg (TU) TSX-011 twice daily OR
  - o Schedule B: 507 mg (TU) TSX-011 once daily.

In this case subjects will be stratified during treatment assignment per their Japanese/non-Japanese ethnicity. All study subjects will be manually assigned to schedule A or B to ensure a balanced dosing schedule.

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

Table 1: Adaptive Design and Dose Adjustment Criteria

| Period 2 - Days 1 to 15 | | Period 3 - Dose Adjustment on Day 16 | | | |
|---|---|---|---|---|---|
| Day 8 T level<br>(ng/dL) | Starting<br>Dose (mg) | Frequency | Dose Change | New Dose (mg) | Frequency |
| <350 | 380 | BID | Increase | 570 | BID |
| 350-499 | 380 | BID | Increase | 443 | BID |
| 500-800 | 380 | BID | No change | 380 | BID |
| | | | Decrease | | |
| >800 | 380 | BID | (treatment assignment 1:1) | 317 | BID |
| | | | Decrease | | |
| >800 | 380 | BID | (treatment assignment 1:1) | 507 | QD |

### 3.5.1.2 Dose Adjustment Period 3 Day 26

- If Period 3 Day 19 (6 hours postdose ± 15 minutes) total testosterone is <350 ng/dL, dose adjust subjects to 570 mg TU dosing thrice daily for their Day 26 dose. Dosing times should be (8 am ± 60 minutes, 8 hours post morning dose ± 15 minutes, and 14 hours post morning dose ± 15 minutes).
- If Period 3 Day 19 (6 hours postdose ± 15 minutes) total testosterone is ≥350 ng/dL and <500 ng/dL, then their Day 26 dose will be as follows:
  - a. Dose adjust subjects on once-daily dosing from 507 mg TU daily to 570 mg TU daily.
  - b. Dose adjust subjects on twice daily dosing as follows:
    - o If dose is 570 mg TU twice daily, increase to 633 mg TU twice daily.
    - o If dose is 443 mg TU twice daily, increase to 507 mg TU twice daily.
    - o If dose is 380 mg TU twice daily, increase to 443 mg TU twice daily.
    - o If dose is 317 mg TU twice daily, increase to 380 mg TU twice daily.

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

- If period 3 Day 19 (6 hours post-dose ± 15 minutes) total testosterone is between 500 and 800 ng/dL inclusive, continue the current dose for their Day 26 dose.
- If Period 3 Day 19 (6 hours postdose ± 15 minutes) total testosterone is >800 ng/dL, their Day 26 dose should be decreased as follows:
  - a. For once-daily dosing subjects change the dose from 507 mg TU daily to 380 mg TU daily.
  - b. For the twice-daily dosing group:
    - o If dose is 570 mg TU twice daily, decrease to 507 mg TU twice daily.
    - o If dose is 443 mg TU twice daily, decrease to 380 mg TU twice daily.
    - o If dose is 380 mg TU twice daily, decrease to 317 mg TU twice daily.
    - o If dose is 317 mg TU twice daily, decrease to 253 mg TU twice daily.

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

Table 2: Adaptive Design and Dose Adjustment Criteria

| Period 3 - Day 16 to 30 | | | Period 3 - Dose Adjustment on Day 26 | | |
|---|---|---|---|---|---|
| Day 19 T level<br>(ng/dL) | Starting Dose (mg) | Frequency | Dose Change | New Dose<br>(mg) | Frequency |
| <350 | all | | Increase | 570 | TID |
| 350-499 | 570 | BID | Increase | 633 | BID |
| 350-499 | 443 | BID | Increase | 507 | BID |
| 350-499 | 380 | BID | Increase | 443 | BID |
| 350-499 | 317 | BID | Increase | 380 | BID |
| 350-499 | 507 | QD | Increase | 570 | QD |
| 500-800 | 570 | BID | No change | 570 | BID |
| 500-800 | 443 | BID | No change | 443 | BID |
| 500-800 | 380 | BID | No change | 380 | BID |
| 500-800 | 317 | BID | No change | 317 | BID |
| 500-800 | 507 | QD | No change | 507 | QD |
| >800 | 570 | BID | Decrease | 507 | BID |
| >800 | 443 | BID | Decrease | 380 | BID |
| >800 | 380 | BID | Decrease | 317 | BID |
| >800 | 317 | BID | Decrease | 253 | BID |
| >800 | 507 | QD | Decrease | 380 | QD |

BID = twice daily; QD = once daily; TID = thrice daily

### 3.6 Meal Administration

Meals and/or snacks will be provided as appropriate (breakfast, lunch, and dinner) on predose days (e.g., Day -1); thereafter, the meal schedule will be as described in the protocol section 13.7.

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

### 3.7 Interim Analysis

Three starting cohorts of 3 subjects each will complete Periods 1, 2, and 3 prior to enrolment of the remaining subjects. For purpose of this protocol 'enrolment' is the subject first dose (i.e., 190 mg fed Day 1). An interim review of TSX-011 safety and efficacy data (including PK data) will occur prior to enrolling the remaining subjects in the study. Any subject in these cohorts who fails to complete all 3 study periods or is determined to be a non-responder will be replaced.

### 4. PAREXEL Study Analysis Variables

### 4.1 Demographic and Background Variables

The following demographic and anthropometric information will be recorded:

- Date of informed consent
- Medical history (including previous and current medical conditions and medications)
- Drug, alcohol, smoking and caffeine use (previous history and current)
- Age calculated as (date of informed consent date of birth)/365.25
- Gender
- Ethnic origin
- Race
- Height (cm)
- Body weight (kg)
- Body mass index (BMI) (kg/m<sup>2</sup>)

### 4.2 Safety Variables

#### 4.2.1 Adverse Events

Adverse event (AE) monitoring will occur from the time consent is obtained until the end of the subject's participation in the study (i.e., the subject has discontinued or completed the study).

### 4.2.2 Clinical Laboratory Tests

Laboratory safety tests for chemistry, hematology and urinalysis will be performed at the following time points:

Period 1: Screening, Day-1, and Day 2; Period 2: Day 2, Day 8, Day 16; Period 3: Day 31.

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

The following safety laboratory parameters will be measured:

### **Serum Chemistry**

- Albumin
- Alkaline phosphatase
- AST
- ALT
- Blood urea nitrogen
- Creatinine
- Creatine kinase
- Lactate dehydrogenase
- Glucose
- Bilirubin (total)\*
- Total protein
- Sodium
- Potassium
- Calcium
- Chloride
- Total cholesterol
- Triglycerides
- Uric acid
- High-density lipoprotein (HDL)
- Low-density lipoprotein (LDL)

### **Hematology**

- Hemoglobin
- Hematocrit
- Total and differential leukocyte count
- Red blood cell count
- Platelet count
- White blood cell count
- HbA1c\*\*

### **Urinalysis**

- pH
- Specific gravity
- Protein
- Glucose
- Ketones
- Nitrite
- Bilirubin

TesoRx Pharma, LLC Final 1.0
Protocol Number TT-018 13 June 2018

- Blood
- Urobilinogen
- Leukocyte esterase
- Microscopic assessment for cells and casts

Microscopic urinalysis will be performed if urinalysis results are abnormal.

### Virology

- HIV test\*\*
- Hepatitis B surface antigen\*\*
- Hepatitis C virus\*\*

### Urine drug screen \*\*\*

- Cocaine
- Cannabinoids
- Alcohol
- Opiates
- Barbiturates
- Amphetamines
- Benzodiazepines

If total bilirubin results are above the upper limits of normal, direct and indirect bilirubin analysis will be performed.

- \*\* To be performed at screening only.
- \*\*\* To be performed at screening and at each confinement check-in.

After screening, safety laboratory tests will be performed in the fasted state (at least 8 hours fasted).

### 4.2.2.1 Other Lab Assessments - Testosterone Levels, PSA

Testosterone levels will be collected at the following times for each treatment period:

Period 1: screening; Day 1, 6 hours post

Period 2: Day 8, 6 hours post

Period 3: Day 19

PSA values will be assessed at screening period 1, Day 31 period 3

### 4.2.3 Vital Signs

Vital signs will be measured and assessed at the following times:

Period 1: Screening, Day-1, on Day 1 at time 0, 6 hours post, 24 hours post;

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

Period 2: Day -1, Day 1 at 0 hour, 8 hours post, 16 hours post; Day 2, Day 8, Day 14, Day 15 at 0 hour, 8 hours post, 16 hours post.

Period 3: Day 16, Day 29, Day 31.

The following vital signs will be measured:

- Blood pressure (systolic and diastolic [mmHg]);
- Pulse (beats per minute [bpm]);
- Oral body temperature (°C);
- Respiratory rate (breaths per minute).

All vital sign measurements will be single measurements.

### 4.2.4 Electrocardiograms

The 12-lead ECGs will be performed at the following times:

Period 1: Screening, Day-1, on Day 2;

Period 2: Day 2, Day 8.

Period 3: Day 16, Day 31.

The following ECG parameters will be collected: PR interval, QRS interval, RR interval, QT interval, and QTc interval (QTcB and QTcF).

The ECG will be evaluated by the Investigator as 'Normal', 'Abnormal, NCS' or 'Abnormal, CS'.

### 4.2.5 Physical Examination

Physical examinations will be performed at the following times for each period:

Period 1: Screening, Day -1, Day 2;

Period 2: Day -1, Day 14;

Period 3: Day 16, Day 29, Day 31.

#### 4.2.6 Concomitant Medications

Concomitant medication use will be recorded for the 30 days prior to Screening until the final discharge visit (i.e., end of the study).

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

### 4.3 Quality of Life Assessments

Measurements of QOL related to hypogonadal symptoms will be assessed at the following time points: Screening; Period 2: Day -1, Day 15; Period 3: Day 19, Day 31. QOL will be assessed by applying the following questionnaires:

- International Prostrate Symptom Score (IPSS)
- AMS scale
- Male Sexual Dysfunction Multinational Survey of the Aging male (MSAM-7, libido questions only)
- Psychosexual Daily Questionnaire (PDQ)

#### 4.4 Pharmacokinetic Variables

**Period 1**: Blood samples for the determination of endogenous testosterone and DHT will be collected for a single 24-hour period before any study subject exposure to TSX-011. This baseline assessment of endogenous testosterone and DHT will be assessed over a 24-hour predose interval (Day -1) at 0, 1.5, 3, 4.5, 6, 8, 12, 16, and 24 hours.

Blood samples for 24-hour post-dosing will be collected on Day 1 of each dosing PK (190, 380, 570 mg TU) at 0, 1.5, 3, 4.5, 6, 8, 12, 16, and 24 hours.

**Period 2:** Blood samples for determination of PK measurements will be collected at 0, 1.5, 3, 4.5, 6, 8, 10, 11.5, 13, 14.5, 16, 18, and 24 hours on Day 1 and Day 15. The three initial cohorts of 3 subjects each will have additional PK samples taken. Specifically, duplicate PK samples (one serum and one plasma) will be taken on Day 8 prior to dosing and at 6 hours (± 15 minutes) after the morning dose.

The plasma sample values will be used to dose adjust according to the adaptive dosing design.

For the first cohort, if TU is detectable at a level 5 times above the LLOQ (i.e. 10 ng/ml) in the previously collected Day 8 samples, then for PK assessments on Day 15, all blood samples will be collected in duplicate (one serum and one plasma).

For the second and third cohorts, Day 15 samples will be collected in duplicate. The serum sample shall be processed initially, and only if TU is detectable at a level 5 times above the LLOQ (i.e. 10 ng/ml) shall the enzyme inhibited plasma sample undergo PK analysis.

TesoRx Pharma, LLC Final 1.0
Protocol Number TT-018 13 June 2018

**Period 3:** On Day 30, PK samples for a 24-hour PK profile will be obtained at the following sampling times based upon the daily dosing regimen.

For subjects on once daily dosing, blood samples for determination of PK measurements will be collected at 0, 1.5, 3, 4.5, 6, 8, 12, 16, and 24 hours.

For subjects on twice daily dosing, blood samples for determination of PK measurements (4-6 mL blood per time point) will be collected at 0, 1.5, 3, 4.5, 6, 8, 10, 11.5, 13, 14.5, 16, 18, and 24 hours.

For subjects on thrice daily dosing, blood samples for PK determination will be collected at 0, 1.5, 3, 4.5, 6, 8, 9.5, 11, 12.5, 14, 15.5, 17, 18.5, 20, and 24 hours.

The three initial cohorts of 3 subjects each will have additional PK samples taken. Specifically, duplicate PK samples (one serum and one plasma) will be taken on Day 19 at 6 hours (± 15 minutes) after the morning dose. The plasma sample values will be used to dose titrate according to the adaptive dosing design.

### **PK Parameters**

Derivation of all PK parameters will be the responsibility of the sponsor.

The following PK parameters will be calculated using both actual testosterone concentrations following dose administration of TSX-011:

AUC<sub>12</sub>: The area under the concentration versus time curve, from time 0 to

the last measurable concentration on or before time 12 hours, as

calculated by a linear trapezoidal method.

AUC<sub>24</sub>: The area under the concentration versus time curve, from time 0 to

the last measurable concentration on or before time 24 hours, as

calculated by a linear trapezoidal method.

C<sub>max</sub>: Maximum measured concentration over the time span specified.

C<sub>avg</sub>: Average measured concentration over the time span specified.

C<sub>min</sub>: Minimum measured concentration over the time span specified.

T<sub>max</sub>: Time of the maximum measured concentration. If the maximum

value occurs at more than one time point, Tmax is defined as the

first time point with this value.

T<sub>min</sub>: Time of the minimum measured concentration.

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

**Table 2: Pharmacokinetic Parameters** 

| Parameter | Definition | Method of Determination |
|---|---|---|
| Cmax | Maximum plasma TSX-011 concentration | Taken directly from bioanalytical data |
| Tmax | The time to reach Cmax | Taken directly from merged clinical and bioanalytical data, with time presented as actual elapsed time relative to dose |

#### 4.4.1 Pharmacokinetic Parameter Calculation Methods

PK parameters will be calculated by non-compartmental analysis methods from the concentration-time data following these guidelines:

- Actual sampling times relative to dosing rather than nominal times will be used in the calculation of all derived PK parameters.
- There will be no imputation of missing data.

### 4.5 Pharmacodynamic Variables

Not applicable

### 4.6 Efficacy Variables

Not applicable

### 4.7 Analysis Populations

### 4.7.1 Safety Population

The Safety population is defined as all randomized subjects who received at least one dose of study drug and have at least one post-baseline safety assessment. Subjects will be included in the analysis according to IP received.

### 4.7.2 Pharmacokinetic Population (PK)

The PK population is defined as all randomized subjects for whom at least one PK parameter of interest can be calculated. In general, on a parameter-by-parameter basis,

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

an individual subject's data may be excluded from analysis if insufficient data are available for that subject to calculate the specific parameter in question.

### 5. STATISTICAL REPORTING

For the purposes of this SAP IP refers to any dose amount of study drug TSX-011.

#### 5.1 General Considerations for Data Presentations

Data for all enrolled subjects will be presented in the data listings.

A subject who is enrolled but does not receive IP will be included in those data listings for which they have data but will be excluded from all data summaries. Data summaries will only include those subjects that receive IP.

For those listings or data summaries where baseline and change from baseline measurements will be presented, unless stated otherwise the last observed measurement prior to the first dose of IP in a given period will be considered the baseline measurement for the post-dose assessments in that period.

All pre- and post-dose assessments, including unscheduled assessments and repeats, will be included in the data listings. For unscheduled (repeat) assessments collected pre-dose, the last assessment taken for a time point will be used in the data summaries (summary tables, figures, and statistical analysis); for all post-dose time points, the original assessment for any given time point will be used in the data summaries (summary tables, figures, and statistical analysis).

For data summaries of continuous variables will be summarized using descriptive statistics including: number of observations (n), mean (arithmetic and/or geometric), median, standard deviation (SD), minimum, and maximum. Frequencies and percentages will be used for summarizing discrete (categorical) data. In summaries for safety the denominator for all percents will be the number of subjects in a given treatment group.

Data that are reported as missing will be excluded from all descriptive and non-descriptive data analysis. There will be no imputation of data. Observations that might be considered spurious (extreme relative to the majority of the data) will not be altered or removed from any presentation of the data, including the calculation of summary statistics (means, medians, etc.), unless approved by the sponsor.

For data listings, all raw data will be reported/displayed exactly as provided. For summaries of quantitative safety data, the minimum and maximum value will be reported exactly as the raw data are reported; measures of central tendency (means,

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

medians) will be reported to one more decimal place than the raw data; measures of variance (SD) will be reported to two more decimal places than the raw data. Methods for summarizing PK data are described in section 7 of this SAP.

Listings will include all subjects and will be sorted by subject number and time point (where applicable). All derived data used in a data summary or statistical analysis will be listed. All data listings will include a column for treatment period and subject number.

#### 5.2 Treatment Identification

The following will be used to identify the treatment in applicable data listings, tables and figures:

### **Period 1 Treatment**

- 190 mg TSX-011, Fed
- 190 mg TSX-011, Fasted
- 380 mg TSX-011, Fed
- 570 mg TSX-011, Fed

Period 2 Treatment: 380 mg TSX-011 BID dosing, Fed

<u>Period 3 Treatment:</u> Treatments to be determined during dose-adjusted adaptive design period. TSX-011 dose adjustment permitted on Day 16 and Day 26 based on 6 hours post-dose (± 15 minutes) testosterone level on Day 8 and Day 19, respectively; dosing period of 15 days. See Table 1 and Table 2 of this SAP.

#### **SOFTWARE**

All statistical analyses performed by PAREXEL will be performed using Statistical Analysis Software (SAS®) (SAS® Institute Inc., Cary, North Carolina, United States of America [USA]) Version 9.2 or higher. The PK analysis will be performed using Phoenix® WinNonlin® Software Version 6.3 or higher (Certara, L.P., 9666 Olive Blvd, Suite 425, St. Louis MO 63132).

### 6. Subject and Treatment Information

### 6.1 Subject Disposition

The completion status, date of completion or discontinuation, the reason for discontinuation, and the date of withdrawal will be listed (Listing 16.2.1). The number of subjects enrolled and the frequency and percentage of subjects completing the

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

study, subjects withdrawing early, and primary reason for withdrawal will be summarized overall subjects enrolled (Table 14.1.1). The number and percent of subjects in the safety population and PK population will be summarized overall subjects enrolled.

### 6.2 Eligibility Criteria and Protocol Deviations

Listing 16.2.2.1 will display all enrolled subjects who did not meet an inclusion criterion and all enrolled subjects who met an exclusion criterion.

All reported protocol deviations will be listed (Listing 16.2.2.2).

#### **6.3 Exclusion Tests**

Results of all exclusion tests (serology, drug, and alcohol screen) will be listed (Listing 16.2.2.3).

### 6.4 Demographic Data

Demographic information will be listed (Listing 16.2.4.1). Descriptive statistics will be obtained for the continuous variables: height, age, BMI, and body weight presented overall subjects enrolled (Tables 14.1.2). Frequencies and percentage of subjects will be tabulated overall subjects enrolled for the categorical variables ethnicity, race, and gender (Tables 14.1.3).

### 6.5 Medical History

Medical history data will be listed for each subject. Medical history will be coded using Medical Dictionary Regulatory Activities (MedDRA Version 20.1). Only those body systems where a condition or abnormality has been reported will be listed (Listing 16.2.4.2).

#### 6.6 Concomitant Medication

Prior and concomitant medications will be listed by subject (Listings 16.2.5.1 and 16.2.5.2, respectively). Medications will be coded using WHODDE version September 2017.

#### 6.7 Dose Administration

Listing 16.2.5.3 will present subject number, treatment, period, visit, and the date and time of dose administration of TSX-011.

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

#### 7. Pharmacokinetic Concentrations and Parameters

Creation and delivery of all pharmacokinetic outputs for concentrations and parameters will be the responsibility of the sponsor.

The PK sample concentrations for all subjects for each period will be summarized for each nominal sample time using minimum, maximum, median, standard deviation, and geometric mean.

The following descriptive statistics will be presented in PK parameter summary tables: n (number of non-missing observations), arithmetic mean, SD, median, minimum, maximum, and geometric mean.

Descriptive statistics and statistical analyses will be calculated using un-rounded results. All PK tables will be presented in units of ng/mL.

#### 7.1 Plasma Concentrations

The minimum and maximum statistics for  $C_{max}$  and summaries of PK concentrations will reflect the rounding shown in the source data as provided by the bioanalytical laboratory.

Pharmacokinetic concentration data for TSX-011 administration will be listed by subject, period, and treatment. Actual sampling times relative to dosing, nominal scheduled times, and the difference between the actual and nominal sample time will also be listed. PK concentrations presented will include only actual total testosterone concentrations.

### 8. Safety Analysis

The analysis of the safety variables will be conducted using the safety population.

#### 8.1 Adverse Events

All verbatim AE terms reported will be coded according to MedDRA, version 20.1.

Adverse events will be categorized as:

- Treatment emergent AEs (TEAEs) are defined as any AEs that occur after first dose of IP
- Non-treatment emergent AEs (NTEAE): AEs whose onset occurred before the administration of first IP

All AE data as captured in ClinBase will be listed for each subject (Listing 16.2.7.1). All serious AEs (SAEs) will be listed (Listing 16.2.7.2). A listing of all AEs leading to treatment discontinuation will be presented, if applicable (Listing 16.2.7.3).

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

Unless specified otherwise, all adverse event summaries will include the TEAEs only and adverse event summary counts of AEs will be the number of subjects reporting adverse events and not the number of events reported. The number and percentage of subjects with adverse events will be tabulated by body system and preferred term by treatment. A subject with multiple adverse events within a body system is only counted once towards the total of that body system. If the same AE (preferred term) is reported several times for the same subject within a given treatment, it will only appear once for that specified treatment in the summary tables.

For purposes of the summary tables, AEs will be classified as either being related to study drug or not related. AEs related to study drug will include AEs classified as 'Definite', 'Probable', or 'Possible'. AEs not related to study drug will include AEs that are 'Not related'.

As defined in the protocol, within the source data all AEs will be assigned a severity grade of: Mild, Moderate, or Severe. For subjects with multiple adverse events of the same preferred term and of different severities, the AE with the highest assessment of severity will be used in the summaries presented by severity.

A general summary of all treatment-emergent adverse events (Table 14.3.1.1) will show the number and percentage of subjects, as well as the number of events, according to the following categories:

- All treatment emergent adverse events
- Treatment emergent adverse events 'Related' to TSX-011
- Mild treatment emergent adverse events
- Moderate treatment emergent adverse events
- Severe treatment emergent adverse events
- Serious treatment emergent adverse events
- Treatment emergent adverse events leading to early termination
- Deaths

Other summary tables for adverse events will include:

- Table 14.3.1.2: Number and Percentage of Subjects with Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Treatment
- Table 14.3.1.3: Number and Percentage of Subjects with Treatment Emergent Adverse Events 'Related to the IP' by System Organ Class, Preferred Term, Severity, and Treatment.
- Table 14.3.1.4: Number and Percentage of Subjects with Treatment Emergent Adverse Events 'Not Related to the IP' by System Organ Class, Preferred Term, Severity, and Treatment.

For tabulations of AEs by treatment, any AE that starts on or after administration of the first dose period 1 (i.e. Period 1, 190 mg fed) and before the second dose period 1

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

(Period 1, 190 mg fasted), will be assigned to the first treatment dose period 1. Any AE occurring after the second dose period 1 (Period 1, 190 mg fasted) and before the third dose period 1 (Period 1, 380 mg), will be assigned to the second dose; and any AE occurring after the third dose period 1 (Period 1, 380 mg) and before the first dose of treatment period 2 (Period 2, 380 mg) will be assigned to the period 1 third dose.

If a subject has multiple AEs with the same preferred term but occurring after each dose administration, then one AE will be counted for each treatment. Adverse events that emerge in one treatment period and carry over into the next period will be attributed to only the period in which the AE emerged.

### 8.2 Clinical Safety Laboratory Tests (Hematology, Chemistry, Urinalysis)

### 8.2.1 Hematology and Chemistry

A by-subject listing of all observed chemistry and hematology laboratory data will be provided (Listings 16.2.8.1 and 16.2.8.2, respectively). Laboratory results outside the normal range will be flagged. The abnormal values will be flagged with 'L' (low) for values below the lower limit of the laboratory's normal range or 'H' (high) for values above the upper limit of the laboratory's normal range. Abnormal values will be graded as not clinically significant (NCS) or clinically significant (CS). Clinically significant laboratory results will be included in the AE listings.

The observed values of all safety laboratory assessments for clinical chemistry and hematology will be summarized using descriptive statistics showing the number of observations (n), mean, median, SD, minimum, and maximum value. Table summaries will be presented overall treatments for each time point: (Chemistry Table 14.3.2.1, Hematology Table 14.3.2.2).

Baseline values for all clinical chemistry and hematology parameters will be categorized as being below the normal range (Low), within the normal range (Normal), and above the normal range (High). Shift from baseline tables will present the frequency and percentage of subjects who have observations that are Normal, Low, or High. Shift tables will be presented by time point overall treatments (Tables 14.3.2.3 and 14.3.2.4). For shift tables, baseline will be the last laboratory assessment prior to the first dose in Period 1.

Only laboratory parameters noted in Section 4.2.2 of this SAP will be tabulated.

### 8.2.2 Urinalysis

Urinalysis test results for pH, specific gravity, protein, glucose, ketones, bilirubin, blood, nitrite, urobilinogen, leukocyte esterase will be listed (Listing 16.2.8.3). All positive findings in the microscopic examination will be listed (Listing 16.2.8.4).

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

Observations outside the normal range will be flagged. The abnormal quantitative values will be flagged with 'L' for values below the lower limit of the laboratory's normal range, 'H' for values above the upper limit of the laboratory's normal range, or 'Ab' for abnormal qualitative test results. All original and unscheduled assessments will be listed. Clinically significant laboratory results that are considered by the investigator to be AEs will be included in the AE listings.

### **8.2.3 Laboratory Comments**

A listing of laboratory comments will be provided (Listing 16.2.8.5).

#### 8.2.4 Other Laboratory Assessments

Results for testosterone and PSA will be listed for each subject.

### 8.3 Vital Signs

The observed data for blood pressure (systolic and diastolic), heart rate (pulse), body temperature and respiration rate will be listed by subject, treatment, and time point (Listings 16.2.9.1). Change from baseline for blood pressure (systolic and diastolic), heart rate (pulse), body temperature and respiration rate will be derived and listed by subject, treatment, and time point (Listing 16.2.9.2).

In the calculation of change from baseline, the baseline value for each period will be the last assessment collected prior to first dosing in each treatment period.

For systolic and diastolic blood pressure, heart rate, body temperature and respiration rate the observed and change from baseline data will be summarized by treatment and time point. Summaries will include tables of descriptive statistics showing the number of observations (n), mean, SD, median, minimum, and maximum value (Tables 14.3.3.1 and 14.3.3.2).

### 8.4 12-Lead Safety ECG

Raw quantitative results for: PR interval, QRS interval, RR interval, QT interval, QTcB (corrected QT according to Bazett), QTcF (corrected QT according to Fridericia), and heart rate will be listed for each subject (Listing 16.2.10.1). Change from baseline will be derived and listed for each subject for parameters QT, QTcB and QTcF (Listing 16.2.10.2).

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

In the calculation of change from baseline, the baseline value for each period will be the last assessment collected prior to first dosing in each treatment period.

The overall qualitative ECG assessment for each subject will be listed by treatment, subject, and time point (Listing 16.2.10.3).

For QT, QTcB, and QTcF the observed and change from baseline data will be summarized by time point. Summaries will include tables of descriptive statistics showing the number of observations (n), mean, SD, median, minimum, and maximum value (Table 14.3.4.1).

The number and percentage of subjects having observed QT, QTcB, and QTcF values that satisfy the following conditions will be summarized by time point (Table 14.3.4.2):

- < 450 msec
- $450 < \text{to} \le 480 \text{ msec}$
- 480 < to < 500 msec
- > 500 msec

The number and percentage of subjects having change from baseline QT, QTcB, and QTcF values that satisfy the following conditions will be presented by time point (Table 14.3.4.3):

- $\leq 0$  msec
- > 0 to < 30 msec
- $> 30 \text{ to} \le 60 \text{ msec}$
- $\bullet$  > 60 msec

### 8.5 Physical Examination

All abnormal physical examination findings (pre and post-dose assessments) will be listed (Listing 16.2.11).

### 8.6 IPSS Questionnaire

Results from the IPS questionnaire will be listed for each subject by treatment period (Listing 16.2.12.1).

### 8.7 QOL Questionnaire

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

Results from the QOL questionnaire will be listed for each subject by treatment period (Listing 16.2.12.2). Including will be results for IPSS, AMS scale, MSAM-7, and PDQ.

### 9. Reporting Output

The tables, listings, figures and any non-descriptive statistical analysis will be produced using Unix SAS® Software (Version 9.0 or higher). The REPORT procedure will be used to produce all tables and listings; SAS/GRAPH will be used to produce all figures.

Tables, listings, and figures will be produced in the order that they appear in the textual sections of the plan.

All tables, listings, and graphs will be produced to landscape orientation using Courier New 8pt font and will be incorporated into a MS Word document as a (RTF) rich text file (margins: top, left, right, and bottom: 1 inch). A separate RTF document will be created for each table, figure and listing individually.

### 10. References

1. Phoenix<sup>®</sup> WinNonlin<sup>®</sup> version 6.3 or higher (Certara, L.P., 9666 Olive Blvd, Suite 425, St. Louis MO 63132).

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

### 11. Summary Tables

| Table 14.1.1 | Subject Disposition |
|----------------|-------------------------------------------------------------|
| Table 14.1.2 | Demographics - Continuous Variables |
| Table 14.1.3 | Demographics - Categorical Variables |
| Table 14.3.1.1 | Summary of Treatment Emergent Adverse Events |
| Table 14.3.1.2 | Number and Percentage of Subjects with Treatment Emergent |
| | Adverse Events by System Organ Class, Preferred Term, and |
| | Treatment |
| Table 14.3.1.3 | Number and Percentage of Subjects with Treatment Emergent |
| | Adverse Events 'Related to the IMP' by System Organ Class, |
| | Preferred Term, Severity, and Treatment |
| Table 14.3.1.4 | Number and Percentage of Subjects with Treatment Emergent |
| | Adverse Events 'Not Related to the IMP' by System Organ |
| | Class, Preferred Term, Severity, and Treatment |
| Table 14.3.2.1 | Clinical Laboratory Chemistry Summary of Observed Values |
| Table 14.3.2.2 | Clinical Laboratory Hematology Summary of Observed Values |
| Table 14.3.2.3 | Clinical Laboratory Chemistry Shift From Baseline to Day 5 |
| Table 14.3.2.4 | Clinical Laboratory Hematology Shift From Baseline to Day 5 |
| Table 14.3.3.1 | Vital Signs Blood Pressure and Heart Rate Summary of |
| | Observed and Values |
| Table 14.3.3.2 | Vital Signs Blood Pressure and Heart Rate Summary of Change |
| | From Baseline Values |
| Table 14.3.4.1 | 12-Lead ECG - Summary of Observed and Change From |
| | Baseline Values |
| Table 14.3.4.2 | 12-Lead ECG – Categorical Summary of Observed Values |
| Table 14.3.4.3 | 12-Lead ECG – Categorical Summary of Change From Baseline |

TesoRx Pharma, LLC Protocol Number TT-018

Final 1.0 13 June 2018

### 12. Listings

| Listing 16.2.1 | Subject Disposition |
|---|---|
| Listing 16.2.2.1 | Enrolled Subjects Who Did Not Meet All Eligibility Criteria |
| Listing 16.2.2.2 | Protocol Deviations |
| Listing 16.2.2.3 | Exclusion Tests |
| Listing 16.2.4.1 | Demographics |
| Listing 16.2.4.2 | Medical History |
| Listing 16.2.5.1 | Prior Medications |
| Listing 16.2.5.1 | Concomitant Medications |
| Listing 16.2.5.3 | Dose Administration |
| Listing 16.2.7.1 | Adverse Events |
| Listing 16.2.7.1 | Serious Adverse Events |
| ŭ | Adverse Events Leading to Discontinuation |
| Listing 16.2.7.3 | |
| Listing 16.2.8.1 | Clinical Laboratory Chemistry – Observed Values |
| Listing 16.2.8.2 | Clinical Laboratory Hematology – Observed Values |
| Listing 16.2.8.3 | Clinical Laboratory Urinalysis – Observed Values |
| Listing 16.2.8.4 | Clinical Laboratory Urinalysis – Positive Microscopic Findings |
| Listing 16.2.8.5 | Clinical Laboratory Comments |
| Listing 16.2.8.6 | Other Clinical Laboratory Results |
| Listing 16.2.9.1 | Vital Signs Observed Values |
| Listing 16.2.9.2 | Vital Signs Change from Baseline |
| Listing 16.2.10.1 | 12 Lead Safety ECG Quantitative Findings |
| Listing 16.2.10.2 | 12 Lead Safety ECG Change From Baseline |
| Listing 16.2.10.3 | 12 Lead Safety ECG – Qualitative Assessment |
| Listing 16.2.11 | Physical Examination Abnormal Findings |
| Listing 16.2.12.1 | QOL questionnaire - International Prostrate Symptom Score (IPSS) |
| Listing 16.2.12.2 | QOL questionnaire – AMS |
| Listing 16.2.12.3 | QOL questionnaire – Male Sexual Dysfunction Multinational Survey of |
| | the Aging male (MSAM-7) |
| Listing 16.2.12.4 | QOL questionnaire – Psychosexual Daily Questionnaire (PDQ) |
Final 1.0 13 June 2018

13. Table Shells

Final 1.0 13 June 2018

Page X of Y

TesoRx Pharma, LLC Protocol Number: TT-018

Table 14.1.1
Subject Disposition

| | Overall<br>N = x |
|-----------------------------|------------------|
| Enrolled | nn (nn.n%) |
| Completed the Study | nn (nn.n%) |
| Discontinued from the Study | nn (nn.n%) |
| Safety Population | nn (nn.n%) |
| Pharmacokinetic Population | nn (nn.n%) |
| Reason for Discontinuation | |
| Adverse Event | nn (nn.n%) |
| Protocol Deviation | nn (nn.n%) |
| Consent Withdrawn | nn (nn.n%) |
| Lost to Follow-Up | nn (nn.n%) |
| Death | nn (nn.n%) |
| Other | nn (nn.n%) |

Final 1.0 13 June 2018

Page X of Y

TesoRx Pharma, LLC Protocol Number: TT-018

Table 14.1.2

Demographics - Continuous Variables

| | Statistic | Overall |
|----------|-----------|---------|
| | | N = x |
| | n | nn |
| | Mean | XX.X |
| Age | SD | XX.XX |
| (years) | Median | XX.X |
| | Min | XX |
| | Max | XX |
| | n | nn |
| | Mean | XX.X |
| Height | SD | XX.XX |
| (cm) | Median | XX.X |
| | Min | XX |
| | Max | XX |
| | n | nn |
| | Mean | XX.X |
| Weight | SD | XX.XX |
| (kg) | Median | XX.X |
| | Min | XX |
| | Max | XX |
| | n | nn |
| | Mean | XX.X |
| BMI | SD | XX.XX |
| (kg/m^2) | Median | XX.X |
| | Min | XX |
| | Max | XX |

Final 1.0 13 June 2018

Page X of Y

TesoRx Pharma, LLC Protocol Number: TT-018

### Table 14.1.3 Demographics - Categorical Variables

| | | verall<br>N = x |
|-------------------------------------------|----|-----------------|
| Ethnicity | | |
| Hispanic/Latino | nn | (nn.n%) |
| Non Hispanic/Latino | nn | (nn.n%) |
| Race | | |
| White | nn | (nn.n%) |
| American Indian/Alaska Native | nn | (nn.n%) |
| Asian | nn | (nn.n%) |
| Native Hawaiian or other Pacific Islander | nn | (nn.n%) |
| Black/African American | nn | (nn.n%) |
| Other | nn | (nn.n%) |
| Gender | | |
| Male | nn | (nn.n%) |

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

| | Treatment | | | | | |
|---|---|---|---|---|---|---|
| · | 190 mg<br>TSX-011<br>Fasted<br>N = x | 190 mg<br>TSX-011<br>Fed<br>N = x | 380 mg<br>TSX-011<br>Fed<br>N = x | 570 mg<br>TSX-011<br>Fed<br>N = x | 380 mg<br>TSX-011<br>BID Fed<br>N = x | Period 3<br>Adaptive-Dose<br>Design<br>Treatment |
| | nn (%) E | nn (%) E | nn (%) E | nn (%) E | nn (%) E | nn (%) E |
| All AEs | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |
| AEs 'Related to TSX-011' | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |
| AEs 'Related to both' | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |
| Mild AEs | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |
| Moderate AEs | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |
| Severe AEs | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |
| Deaths | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |
| Serious AEs | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |
| AEs Leading to discontinuation of IMP | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E | nn (nn.n%) E |

TEAE = Treatment Emergent Adverse Event nn = Number of Subjects with TEAEs N = Number of Subjects Exposed (nn.n%) = nn/N x 100

E = Number of AEs

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Table 14.3.1.2

Number and Percentage of Subjects with Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Treatment

| | | Treatment | | | | |
|---|---|---|---|---|---|---|
| System Organ Class Preferred Term | 190 mg<br>TSX-011<br>Fasted | 190 mg<br>TSX-011<br>Fed | 380 mg<br>TSX-011<br>Fed | 570 mg<br>TSX-011<br>Fed | 380 mg<br>TSX-011<br>BID Fed | Period 3<br>Adaptive-<br>Dose |
| ricicited icim | N = x | N = x | N = x | N = x | N = x | Design<br>Treatment |
| System Organ Class 1 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 1 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 2 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 3 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term xx | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| System Organ Class 2 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 1 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 2 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 3 | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term xx | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018 Page X of Y

Table 14.3.1.3

Number and Percentage of Subjects with Treatment Emergent Adverse Events 'Related to IP' by System Organ Class, Preferred Term, Severity, and Treatment

| | | | | Treatme | ent | | |
|---|---|---|---|---|---|---|---|
| | _ | 190 mg | 190 mg | 380 mg | 570 mg | 380 mg | Period 3 |
| System Organ Class | | TSX-011 | TSX-011 | TSX-011 | TSX-011 | TSX-011 | Adaptive- |
| Preferred Term | Severity | Fasted | Fed | Fed | Fed | BID Fed | Dose |
| 110101100 101 | 55.02201 | N = X | N = x | N = X | N = x | N = x | Design |
| | | | | | | | Treatment |
| System Organ Class 1 | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 1 | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term xx | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| System Organ Class 2 | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term 1 | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Preferred Term xx | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) |
| Etc | | | | | | | |

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Table 14.3.1.4

Number and Percentage of Subjects with Treatment Emergent Adverse Events 'Not Related to IP' by System Organ Class, Preferred Term, Severity, and Treatment

| | | | | Treatme | ent | | |
|---|---|---|---|---|---|---|---|
| | _ | 190 mg | 190 mg | 380 mg | 570 mg | 380 mg | Period 3 |
| Q.,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | | TSX-011 | TSX-011 | TSX-011 | TSX-011 | TSX-011 | Adaptive- |
| System Organ Class | G ! b | Fasted | Fed | Fed | Fed | BID Fed | Dose |
| Preferred Term | Severity | N = x | N = x | N = X | N = X | N = x | Design |
| | | | | | | | Treatment |
| System Organ Class 1 | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| Preferred Term 1 | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| Preferred Term xx | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| System Organ Class 2 | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| Preferred Term 1 | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| Preferred Term xx | Mild | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| | Moderate | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |
| | Severe | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n%) | nn (nn.n% |

Final 1.0 13 June 2018

Page X of Y

TesoRx Pharma, LLC Protocol Number: TT-018

Table 14.3.2.1 Clinical Laboratory Chemistry - Summary of Observed Values

| | | Overall |
|-----------|-----------|---------|
| Visit | Statistic | N = x |
| | n | nn |
| | Mean | XX.X |
| Screening | SD | XX.XX |
| | Median | XX.X |
| | Min | XX |
| | Max | XX |
| | n | nn |
| | Mean | XX.X |
| | SD | xx.xx |
| Day -1 | Median | XX.X |
| | Min | XX |
| | Max | xx |
| | n | nn |
| | Mean | XX.X |
| Day 2 | SD | XX.XX |
| Day Z | Median | XX.X |
| | Min | XX |
| | Max | XX |
| | n | nn |
| | Mean | XX.X |
| Day 2 | SD | XX.XX |
| 2 | Median | XX.X |
| Period 2 | Min | XX |
| | Max | XX |
| | n<br>Moan | nn<br> |
| Da 0 | Mean | XX.X |
| Day 8 | SD | XX.XX |
| Danial O | Median | XX.X |
| Period 2 | Min | XX |
| E+ o | Max | XX |
| Etc | | |

Final 1.0 13 June 2018

Page X of Y

TesoRx Pharma, LLC Protocol Number: TT-018

Table 14.3.2.2 Clinical Laboratory Hematology - Summary of Observed Values

| | | Overall |
|-----------|-----------|---------|
| Visit | Statistic | N = x |
| | n | nn |
| | Mean | XX.X |
| Screening | SD | XX.XX |
| | Median | XX.X |
| | Min | XX |
| | Max | XX |
| | n | nn |
| | Mean | xx.x |
| | SD | XX.XX |
| Day -1 | Median | XX.X |
| | Min | XX |
| | Max | XX |
| | n | nn |
| | Mean | XX.X |
| Day 2 | SD | XX.XX |
| Day 2 | Median | XX.X |
| | Min | XX |
| | Max | XX |
| | n | nn |
| | Mean | XX.X |
| Day 2 | SD | xx.xx |
| - | Median | XX.X |
| Period 2 | Min | xx |
| | Max | XX |
| | n | nn |
| | Mean | XX.X |
| Day 8 | SD | XX.XX |
| Day 0 | Median | XX.X |
| Period 2 | Min | XX.X |
| 101100 2 | Max | XX |
| | 1147 | AA |

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Table 14.3.2.3.1 Clinical Laboratory Chemistry - Shift From Baseline to Maximum Value Post-Dose

| | | | Baseline (Day -1) | | | | |
|---|---|---|---|---|---|---|---|
| | Shift | | Low | 1 | Normal | | High |
| Treatment | From | | | | | | |
| Period | Baseline | | | | | | |
| Period 1 | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| Period 2 | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| Period 3 | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |

Final 1.0 13 June 2018

Page X of Y

TesoRx Pharma, LLC Protocol Number: TT-018

Table 14.3.2.3.2 Clinical Laboratory Chemistry - Shift From Baseline to Minimum Value Post-Dose

| | | Baseline (Day -1) | | | | | |
|---|---|---|---|---|---|---|---|
| | Shift | | Low | 1 | Normal | | High |
| Treatment | From | | | | | | |
| Period | Baseline | | | | | | |
| Period 1 | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| Period 2 | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| Period 3 | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | 2 | | | | | | |

Final 1.0 13 June 2018

Page X of Y

TesoRx Pharma, LLC Protocol Number: TT-018

 ${\tt Table~14.3.2.4.1} \\ {\tt Clinical~Laboratory~Hematology~-~Shift~From~Baseline~to~Maximum~Value~Post-Dose} \\$ 

| | | Baseline (Day -1) | | | | | |
|---|---|---|---|---|---|---|---|
| | Shift | | Low | 1 | Normal | | High |
| Treatment | From | | | | | | |
| Period | Baseline | | | | | | |
| Period 1 | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| Period 2 | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| Period 3 | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |

Final 1.0 13 June 2018

Page X of Y

TesoRx Pharma, LLC Protocol Number: TT-018

 ${\tt Table~14.3.2.4.2} \\ {\tt Clinical~Laboratory~Hematology~-~Shift~From~Baseline~to~Minimum~Value~Post-Dose} \\$ 

| | | | Baseline (Day -1) | | | | |
|---|---|---|---|---|---|---|---|
| | Shift | | Low | 1 | Normal | | High |
| Treatment | From | | | | | | |
| Period | Baseline | | | | | | |
| Period 1 | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | Low | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| Period 2 | Normal | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |
| Period 3 | Low<br>Normal | nn<br>nn | (nn.n%)<br>(nn.n%) | nn<br>nn | (nn.n%)<br>(nn.n%) | nn<br>nn | (nn.n%)<br>(nn.n%) |
| reliou 3 | High | nn | (nn.n%) | nn | (nn.n%) | nn | (nn.n%) |

Final 1.0 13 June 2018

Page X of Y

TesoRx Pharma, LLC Protocol Number: TT-018

Table 14.3.3.1
Vital Signs Summary of Observed Values

#### Parameter = Systolic Blood Pressure (mmHg)

| | | Overall<br>N = x |
|---|---|---|
| Visit | Statistic | N - X |
| Screening | n<br>Mean<br>SD<br>Median<br>Min<br>Max | nn<br>xx.x<br>xx.xx<br>xx.x<br>xx.x<br>xx |
| Day -1 | n<br>Mean<br>SD<br>Median<br>Min<br>Max | nn<br>xx.x<br>xx.xx<br>xx.x<br>xx.x<br>xx |
| Day 1,<br>Time 0 | n<br>Mean<br>SD<br>Median<br>Min<br>Max | nn<br>xx.x<br>xx.xx<br>xx.x<br>xx.x |
| Day 1, 6 hours post | n<br>Mean<br>SD<br>Median<br>Min<br>Max | nn<br>xx.x<br>xx.xx<br>xx.x<br>xx |

Final 1.0 13 June 2018

Page X of Y

TesoRx Pharma, LLC Protocol Number: TT-018

Table 14.3.3.2
Vital Signs Summary of Change from Baseline

Parameter = Systolic Blood Pressure (mmHg)

| Visit | Statistic | Overall<br>N = x |
|---|---|---|
| Day 1, 6<br>hours<br>post | n<br>Mean<br>SD<br>Median<br>Min<br>Max | nn<br>xx.x<br>xx.xx<br>xx.x<br>xx<br>xx |
| Day 1, 24<br>hours<br>post | n<br>Mean<br>SD<br>Median<br>Min<br>Max | nn<br>xx.x<br>xx.xx<br>xx.x<br>xx.x<br>xx |
| Period 2,<br>Day 1, 8<br>hours<br>post | n<br>Mean<br>SD<br>Median<br>Min<br>Max | nn<br>xx.x<br>xx.xx<br>xx.x<br>xx |
| Period 2,<br>Day 1, 16<br>hours<br>post | n<br>Mean<br>SD<br>Median<br>Min<br>Max | nn<br>xx.x<br>xx.xx<br>xx.x<br>xx<br>xx |

Baseline in a given period is the last assessment prior to the first dose in that period.

Final 1.0 13 June 2018

Page X of Y

TesoRx Pharma, LLC Protocol Number: TT-018

Table 14.3.4.1
12 Lead ECG - Summary of Observed and Change From Baseline Values

Parameter = QT (msec)

| | | Observed | Change From |
|-----------|-----------|----------|-------------|
| | | | Baseline |
| Visit | Statistic | N = x | N = x |
| | n | nn | |
| | Mean | XX.X | |
| Screening | SD | XX.XX | |
| | Median | XX.X | |
| | Min | XX | |
| | Max | XX | |
| | n | nn | |
| | Mean | XX.X | |
| Day -1 | SD | XX.XX | |
| | Median | XX.X | |
| | Min | XX | |
| | Max | XX | |
| | n | nn | nn |
| | Mean | XX.X | XX.X |
| Day 2 | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Min | XX | XX |
| | Max | XX | XX |
| | n | nn | nn |
| | Mean | XX.X | XX.X |
| Period 2 | SD | XX.XX | XX.XX |
| Day 2 | Median | XX.X | XX.X |
| | Min | XX | XX |
| | Max | XX | XX |
| Etc | | | |

Baseline = Day -1

QTcB = QT corrected according to Bazett, QTcF = QT corrected according to Fridericia.

Programming Notes: Table will be expanded to include QT, QTcB, and QTcF

Final 1.0 13 June 2018

Page X of Y

TesoRx Pharma, LLC Protocol Number: TT-018

Table 14.3.4.2
12 Lead ECG - Categorical Summary of Observed Values

Parameter = QT (msec)

| | | Overall |
|-----------|--------------------|------------|
| Visit | Category (unit) | |
| | | N = x |
| | ≤ 450 | nn (nn.n%) |
| Screening | $450 < to \le 480$ | nn (nn.n%) |
| screening | $480 < to \le 500$ | nn (nn.n%) |
| | >500 | nn (nn.n%) |
| | ≤ 450 | nn (nn.n%) |
| Day -1 | $450 < to \le 480$ | nn (nn.n%) |
| _ | $480 < to \le 500$ | nn (nn.n%) |
| | >500 | nn (nn.n%) |
| | ≤ 450 | nn (nn.n%) |
| | $450 < to \le 480$ | nn (nn.n%) |
| Day 2 | $480 < to \le 500$ | nn (nn.n%) |
| | >500 | nn (nn.n%) |
| Etc | | |

QTcB = QT corrected according to Bazett, QTcF = QT corrected according to Fridericia.

Programming Notes:

Table will be expanded to include QT, QTcB, and QTcF

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018 Page X of Y

#### 

Parameter = QT (msec)

| | | Overall |
|----------------|--------------------------|------------|
| Visit | Category (unit) | |
| | | N = x |
| | <= 0 | nn (nn.n%) |
| Da.: 2 | >0 to ≤ 30 | nn (nn.n%) |
| Day 2 | >30 to ≤ 60 | nn (nn.n%) |
| | >60 | nn (nn.n%) |
| | <= 0 | nn (nn.n%) |
| | >0 to ≤ 30 | nn (nn.n%) |
| Period 2 Day 2 | >30 to ≤ 60 | nn (nn.n%) |
| | >60 | nn (nn.n%) |
| | <= 0 | nn (nn.n%) |
| | $>0$ to $\leq 30$ | nn (nn.n%) |
| | $>30 \text{ to} \leq 60$ | nn (nn.n%) |
| | >60 | nn (nn.n%) |
| Period 2 Day 8 | | |
| _ | <= 0 | nn (nn.n%) |
| | >0 to ≤ 30 | nn (nn.n%) |
| | >30 to ≤ 60 | nn (nn.n%) |
| | >60 | nn (nn.n%) |

Baseline = Day -1 QTcB = QT corrected according to Bazett, QTcF = QT corrected according to Fridericia.

Programming Notes:
Table will be expanded to include QT, QTcB, and QTcF

Final 1.0 13 June 2018

14. Listing Shells

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018 Page X of Y

Listing 16.2.1 Subject Disposition

If Discontinued, Reason For Period Study Day Subject Completion Status Date of Withdrawal Discontinuation of Withdrawal of Withdrawal Completed

Discontinued

Final 1.0 13 June 2018

Page X of Y

TesoRx Pharma, LLC Protocol Number: TT-018

Listing 16.2.2.1 Enrolled Subjects Who Did Not Meet All Eligibility Criteria

Subject Criteria Category Criteria Description Response

Inclusion No
Exclusion Yes

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.2.2 Protocol Deviations

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.2.3 Exclusion Tests Serology, Drug, Alcohol Screen

Collection Collection Subject Period Visit Date Time Exclusion Test Result

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.4.1 Demographics

Age Height Weight BMI Subject Gender Ethnicity Race (yrs) (cm) (kg) (kg/m^2)

Final 1.0 13 June 2018

Page X of Y TesoRx Pharma, LLC Protocol Number: TT-018

> Listing 16.2.4.2 Medical History

Body System >MedDRA Preferred Term Condition or Date of Date of >>System Organ Class Resolution Subject Abnormality Remark Onset Status

Chronic

Final 1.0 13 June 2018

Page X of Y

TesoRx Pharma, LLC Protocol Number: TT-018

Start Date

Subject

Listing 16.2.5.1

Prior Medications Medications Taken 30 Days Prior to Screening until First Dose of Study Medication

Stop Medication

Dose (units)

Ongoing?

Date

Reason for use

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.5.2 Concomitant Medications

| | | | | | Start | Stop | |
|---|---|---|---|---|---|---|---|
| | | Total dose / | | | Date | Date | Reason |
| Subject | Medication | administration | Route | Frequency | Time | Time | for use |

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.5.3 Study Drug Administration

Date of Time of Drug Dose Dose Dose Subject Treatment Visit Administered Unit Frequency Period Dose Dose Name

Final 1.0 13 June 2018

TesoRx Pharma, LLC
Protocol Number: TT-018

Listing 16.2.7.1 Adverse Events

| | | | | | | | | | | | Time |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | Rela- | | | relative |
| | | | Adverse Event | Start | Stop | | | tion- | Seri- | | to most |
| | | | >MedDRA Preferred Term | Date | Date | | Action | ship | ous | Out- | recent |
| Subject | Period | Treatment | >>Svstem Organ Class | Time | Time | Severity | Taken | to IP | | come | dose |

Final 1.0 13 June 2018

TesoRx Pharma, LLC
Protocol Number: TT-018

Listing 16.2.7.2 Serious Adverse Events

| | | | | | | | | | | Time |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | Rela- | | relative |
| | | | Adverse Event | Start | Stop | | | tion- | | to most |
| | | | >MedDRA Preferred Term | Date | Date | | Action | ship | Out- | recent |
| Subject | Period | Treatment | >>System Organ Class | Time | Time | Severity | Taken | to IP | come | dose |

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.7.3
Adverse Events Leading To Discontinuation

| | | | | | | | | | | | Time |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | Rela- | | | relative |
| | | | Adverse Event | Start | Stop | | | tion- | | | to most |
| | | | >MedDRA Preferred Term | Date | Date | | Action | ship | Seri- | Out- | recent |
| Subject | Period | Treatment | >>Svstem Organ Class | Time | Time | Severity | Taken | to IP | ous | come | dose |

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.8.1 Clinical Laboratory Chemistry - Observed Values

| | Subject | Period | Treatment | Visit | Collection<br>Time | Lab<br>Parameter 1<br>(unit) | Lab<br>parameter 2<br>(unit) | Lab parameter 3 (unit) | Lab parameter 4 (unit) |
|---|---|---|---|---|---|---|---|---|---|
| _ | | | | | | Result/Flag | Result/Flag | Result/Flag | Result/ <i>Flag</i> |

H=High, L=Low, CS=Clinically Significant, NCS=Not Clinically Significant

Programming Note: If Flag is present (H or L), clinical significance will be identified by 'NCS' or 'CS'.

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.8.2 Clinical Laboratory Hematology - Observed Values

| Subject | Period | Treatment | Visit | Collection<br>Time | Lab<br>Parameter 1<br>(unit) | Lab<br>parameter 2<br>(unit) | Lab<br>parameter 3<br>(unit) | Lab<br>parameter 4<br>(unit) |
|---|---|---|---|---|---|---|---|---|
| | | | | | Result/Flag | Result/Flag | Result/Flag | Result/Flag |

H=High, L=Low, CS=Clinically Significant, NCS=Not Clinically Significant

Programming Note: If Flag is present (H or L), clinical significance will be identified by 'NCS' or 'CS'.

Final 1.0 13 June 2018

TesoRx Pharma, LLC Page X of Y

Protocol Number: TT-018

Listing 16.2.8.3
Clinical Laboratory Urinalysis - Observed Values

| | | | | | | Lab | Lab | Lab | Lab |
|---|---|---|---|---|---|---|---|---|---|
| | | | | Collection | Collection | Parameter 1 | parameter 2 | parameter 3 | parameter 4 |
| Subject | Period | Treatment | Visit | Date | Time | (unit) | (unit) | (unit) | (unit) |
| | | | | | | Result/Flag | Result/Flag | Result/Flag | Result/Flag |

H=High, L=Low, AB=Abnormal, CS=Clinically Significant, NCS=Not Clinically Significant

Programming Note: If Flag is present (H, L, or AB), clinical significance will be identified by 'NCS' or 'CS'.

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.8.4 Clinical Laboratory Urinalysis - Positive Microscopic Findings

| | | | | Collection | Collection | | | | | Clinical |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Period | Treatment | Visit | Date | Time | Test Name | Result | Unit | Flag | Significance |

H=High, L=Low, AB=Abnormal, CS=Clinically Significant, NCS=Not Clinically Significant

Programming Note: If Flag is present (H, L, or AB), clinical significance will be identified by 'NCS' or 'CS'.
Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.8.5 Clinical Laboratory Comments

Collection Collection Subject Period Visit Date Time Lab Category Test Name Comment

Lisiting only presents comments associated with our of range results for hematology, chemistry, or urinalysis lab tests.

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.8.6
Other Clinical Laboratory Assessments - Testosterone Levels, PSA

Subject Period Treatment Visit Date Time Lab Lab parameter 2

Result/Flag Result/Flag

H=High, L=Low, AB=Abnormal, CS=Clinically Significant, NCS=Not Clinically Significant

Programming Note: If Flag is present (H, L, or AB), clinical significance will be identified by 'NCS' or 'CS'.

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018 Page X of Y

Listing 16.2.9.1 Vital Signs - Observed Values

| | | | | | | | Diastolic | | Respiratory | Oral |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Systolic Blood | Blood | | Rate | Temperature |
| Subject | | | | Collection | Collection | Pressure | Pressure | Heart Rate | (breaths/min) | (°C) |
| | Period | Treatment | Visit | Date | Time | (mmHg) | (mmHg) | (beats/min) | | |

Final 1.0 13 June 2018

Page X of Y

TesoRx Pharma, LLC
Protocol Number: TT-018

Listing 16.2.9.2 Vital Signs - Change From Baseline

Diastolic Systolic Blood Blood Subject Collection Collection Pressure Pressure Heart Rate (mmHg) Period Treatment Visit Date Time (mmHg) (beats/min)

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.10.1
12 Lead ECG Quantitative Findings

| | | | | | | Heart | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Rate | | | | | | |
| | | | | | | (beats/ | PR | RR | QRS | QT | QTcB | QTcF |
| Subject | Period | Treatment | Visit | Date | Time | min | (msec) | (msec) | (msec) | (msec) | (msec) | (msec) |

QTcB = QT corrected according to Bazett, QTcF = QT corrected according to Fridericia.

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.10.2

12 Lead ECG Quantitative Findings - Change From Baseline

Subject Period Treatment Visit Date Time (msec) (msec) (msec)

QTcB = QT corrected according to Bazett, QTcF = QT corrected according to Fridericia.

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.10.3
12 Lead ECG - Qualitative Assessment

| | | | | Date | Time | | |
|---|---|---|---|---|---|---|---|
| Subject | Period | Treatment | Visit | Taken | Taken | Assessment | Interpretation |
| | | | | | | NORMAL | _ |

ABNORMAL, NCS

NCS = Not Clinically Significant, CS = Clinically Significant

Final 1.0 13 June 2018

TesoRx Pharma, LLC
Protocol Number: TT-018

Page X of Y

Listing 16.2.11
Physical Examination Abnormal Findings

| Subject | Period | Treatment | Visit | Exam<br>Date | Exam<br>Time | Body System | Abnormal<br>Findings | Clinical<br>Significance |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | | NCS<br>CS |

NCS = Not Clinically Significant, CS = Clinically Significant

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.12.1

QOL questionnaire - International Prostrate Symptom Score (IPSS)

| Subject | Period | Treatment | Visit | Date | Time | Symptom | Result | Score |
|---|---|---|---|---|---|---|---|---|
| | | | | | | Incomplete emptying | | |
| | | | | | | Frequency | | |
| | | | | | | Intermittency | | |
| | | | | | | Urgency | | |
| | | | | | | Weak Stream | | |
| | | | | | | Straining | | |
| | | | | | | Nocturia | | |
| | | | | | | Total | | |
| | | | | | | QOL due to Urinary | | |
| | | | | | | Symptoms | | |

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.12.2 QOL questionnaire - AMS

Subject Period Treatment Visit Date Time Symptom Result Score

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.12.3

QOL questionnaire - Male Sexual Dysfunction Multinational Survey of the Aging male (MSAM-7)

Subject Period Treatment Visit Date Time Question Result Score

Final 1.0 13 June 2018

TesoRx Pharma, LLC Protocol Number: TT-018

Page X of Y

Listing 16.2.12.4 QOL questionnaire - Psychosexual Daily Questionnaire (PDQ)

Subject Period Treatment Visit Date Time Question Result Score